CLINICAL TRIAL: NCT00090740
Title: Genetic Risk Factors for Severe Asthma
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: DAIT P01 AI50516
Record Dates: First submitted 2004-09-03; First posted 2004-09-06 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — 40 mL blood

GROUPS / COHORTS (2):
- Asthmatics: People who have asthma
- Controls: People who do not have asthma

SUMMARY:
The purpose of this study is to determine whether a specific genetic factor influences the severity of asthma symptoms.

DETAILED DESCRIPTION:
Asthma is one of the most common chronic diseases in the United States. It is well known that asthma susceptibility is inherited; however, it is unknown if asthma severity is heritable. Studies suggest that levels of interleukin-16 (IL-16) may influence asthma severity. This study will examine the role of differences in the control region of the IL-16 gene in a racially diverse group of asthmatics and nonasthmatics and will determine if the IL-16 gene control region is related to asthma severity.

Participants in this study will undergo lung function and blood tests; they will also complete a questionnaire about their respiratory health. Asthmatic participants will complete a severity-of-asthma questionnaire.

ELIGIBILITY:
Inclusion Criteria for Asthmatic Participants:

* Diagnosis of asthma

Inclusion Criteria for Non-asthmatic Participants:

* No diagnosis of asthma

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 400 asthmatics and 200 non-asthmatic controls will be recruited. The 200 non-asthmatics will be matched for age, gender and ethnicity with the asthmatics in the more severe half of the severity distribution. The participants will be from minority populations (at least 30% African-American and at least 30% Hispanic) and generally of lower socioeconomic status.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2004-09; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Examination of the relationship between the IL-16 promoter genotype and the presence of the asthma phenotype | Throughout study
Examination of the relationship between the IL-16 promoter genotype and asthma severity | Throughout study
Examination of the serum IL-16 concentration and the serum IL-16:IL-9, IL-16:IL-13, and IL-16: TNF-alpha ratios as possible intermediate phenotypes lining the IL-16 promoter genotype to asthma severity | Throughout study

SECONDARY OUTCOMES:
Storage of DNA from all 600 participants for future study into the determinants of asthma severity | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: George O'Connor, MD, Principal Investigator
Locations (1):
- Boston University School of Medicine, Boston, Massachusetts, United States

REFERENCES:
- [Background] Sandford AJ, Chagani T, Zhu S, Weir TD, Bai TR, Spinelli JJ, Fitzgerald JM, Behbehani NA, Tan WC, Pare PD. Polymorphisms in the IL4, IL4RA, and FCERIB genes and asthma severity. J Allergy Clin Immunol. 2000 Jul;106(1 Pt 1):135-40. doi: 10.1067/mai.2000.107926. PMID 10887316
- [Background] Xu J, Meyers DA, Ober C, Blumenthal MN, Mellen B, Barnes KC, King RA, Lester LA, Howard TD, Solway J, Langefeld CD, Beaty TH, Rich SS, Bleecker ER, Cox NJ; Collaborative Study on the Genetics of Asthma. Genomewide screen and identification of gene-gene interactions for asthma-susceptibility loci in three U.S. populations: collaborative study on the genetics of asthma. Am J Hum Genet. 2001 Jun;68(6):1437-46. doi: 10.1086/320589. Epub 2001 May 10. PMID 11349227
- [Background] Lee SY, Lee YH, Shin C, Shim JJ, Kang KH, Yoo SH, In KH. Association of asthma severity and bronchial hyperresponsiveness with a polymorphism in the cytotoxic T-lymphocyte antigen-4 gene. Chest. 2002 Jul;122(1):171-6. doi: 10.1378/chest.122.1.171. PMID 12114354
- [Background] Szalai C, Kozma GT, Nagy A, Bojszko A, Krikovszky D, Szabo T, Falus A. Polymorphism in the gene regulatory region of MCP-1 is associated with asthma susceptibility and severity. J Allergy Clin Immunol. 2001 Sep;108(3):375-81. doi: 10.1067/mai.2001.117930. PMID 11544456